CLINICAL TRIAL: NCT06636409
Title: Long-term Mortality Post Liver Transplantation in the Era of Modern Immunosuppression.
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0432
Record Dates: First submitted 2024-10-02; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Liver Transplant
Keywords: Mortality; Risk factors; Decompensated chronic liver diseases; Survival; Immunosuppression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Liver transplant patients: Liver transplant patients from all French centers between 2008 and 2013 and followed up during the period 2008-2023.
  Interventions: Other: Collection of medical data

INTERVENTIONS:
Other: Collection of medical data — A randomised selection of files to be analyzed will be conducted in each center to constitute a representative sample of liver transplanted patients. This represents 20% of the number of transplanted patients over the period 2008-2013 in the center, allowing a more in-depth analysis of the patients' medical records.

SUMMARY:
Liver transplantation is the primary intervention for decompensated chronic liver diseases and some cases of hepatocellular carcinoma. This study aims to examine long-term mortality after liver transplantation and identify related risk factors in the modern immunosuppression era, using a French multicenter cohort. This study does not interfere with patients' medical care. The study method involves collecting and analyzing only the essential data from patient records.

DETAILED DESCRIPTION:
Liver transplantation stands as the gold standard for treating decompensated chronic liver diseases and select cases of hepatocellular carcinoma. Over time, post-transplant survival rates have shown consistent improvement, attributed to advancements in surgical techniques, refined immunosuppressive protocols, and enhanced comprehension of post-transplant complications. These developments have significantly mitigated the incidence of infectious, immunological, and neoplastic complications following transplantation.

Research indicates post-liver transplant survival rates of approximately 85% at one year, 68% at five years, and 50% at ten years. It is important to note that these statistics are based on patients transplanted in the 1990s, whose immunosuppression relied on a combination of cyclosporine, azathioprine, and corticosteroids.

The field of immunosuppression has undergone substantial evolution, with an expansion in therapeutic options. These include the gradual replacement of Cyclosporine A with Tacrolimus, and the introduction of interleukin-2 receptor inhibitors, mycophenolate mofetil, and mTOR inhibitors. These innovations facilitate more adaptable protocols, offering improved preservation of renal function and allowing for earlier discontinuation of corticosteroids. As a result, these new therapeutic options offer immunosuppression that is more tailored to each patient, with reduced long-term toxicity.

The primary objective of this study is to investigate long-term mortality rates following liver transplantation and to identify the various risk factors contributing to mortality in these patients, with a particular focus on the current era of immunosuppression techniques. This investigation will be conducted within the framework of a French multicentric cohort study.

The results of this study have the potential to enhance our understanding of long-term post-transplant mortality and to more accurately identify risk factors. This knowledge could inform the refinement of immunosuppressive treatments and post-transplant patient care protocols. The overarching aim of this research is to optimize the management of liver transplant recipients and ultimately prolong their survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver transplant between 2008 and 2013 and follow up during 2008-2023

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had liver transplant between 2008 and 2013
Sampling Method: Non-Probability Sample
Enrollment: 1343 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Long-term mortality rates | 1 year, 5 years, and 10 years post-transplant, as well as at the last follow-up
  Evaluation of overall mortality rates among liver transplant recipients, measured from the time of transplantation until the end of the follow-up period.
Risk factors for mortality | 1 year, 5 years, and 10 years post-transplant, as well as at the last follow-up
  Identification of pre- and post-transplant risk factors associated with long-term mortality in liver transplant recipients. Risk factors include demographics (age, sex), comorbidities (diabetes, hypertension, cardiovascular diseases), and transplant-specific factors (MELD score, graft function).

SECONDARY OUTCOMES:
Demographic analysis of transplant recipients | Baseline demographic analysis at 1 year, 5 years, and 10 years post-transplant, as well as at the last follow-up
  Analysis of the demographic characteristics (age, gender, BMI, lifestyle factors such as diabetes, cardiovascular diseases, dyslipidemia, tobacco/alcohol use) of transplant recipients between 2008 and 2013 to determine trends and associations with outcomes
Factors influencing mortality rates | 1 year, 5 years, and 10 years post-transplant, as well as at the last follow-up
  Investigation of specific factors contributing to mortality rates, such as pre-existing liver disease, metabolic conditions and immunosuppressive therapy, in liver transplant recipients
Progression of mortality risk factors | 1 year, 5 years, and 10 years post-transplant, as well as at the last follow-up
  Measurement of how mortality risk factors evolve over time after liver transplantation, focusing on conditions like diabetes, hypertension, renal dysfunction, cardiovascular diseases and graft complications
Mortality rates | 1 year and 5 years post-transplant
  Assessment of mortality rates specifically at the 1-year and 5-year post-transplant milestones to evaluate early and mid-term survival outcomes.
Liver transplant-specific risk factors | 1 year, 5 years, and 10 years post-transplant, as well as at the last follow-up
  Determination of transplant-specific risk factors, including graft rejection, graft dysfunction, recurrence of primary liver disease, and the need for re-transplantation, associated with post-transplant mortality
Non-hepatic risk factors for mortality | 1 year, 5 years, and 10 years post-transplant, as well as at the last follow-up
  Assessment of non-hepatic risk factors associated with post-transplant mortality, encompassing metabolic conditions (such as obesity, hypertension, and diabetes), cardiovascular and renal complications, extra-hepatic malignancies, and infectious diseases

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena MESZAROS, MD, Principal Investigator — Saint Eloi-Hospital, Montpellier
Locations (1):
- Saint Eloi, CHU de Montpellier, Montpellier, France

REFERENCES:
- [Result] Watt KD, Pedersen RA, Kremers WK, Heimbach JK, Charlton MR. Evolution of causes and risk factors for mortality post-liver transplant: results of the NIDDK long-term follow-up study. Am J Transplant. 2010 Jun;10(6):1420-7. doi: 10.1111/j.1600-6143.2010.03126.x. Epub 2010 May 10. PMID 20486907
- [Result] Dopazo C, Bilbao I, Castells LL, Sapisochin G, Moreiras C, Campos-Varela I, Echeverri J, Caralt M, Lazaro JL, Charco R. Analysis of adult 20-year survivors after liver transplantation. Hepatol Int. 2015 Jul;9(3):461-70. doi: 10.1007/s12072-014-9577-x. Epub 2014 Sep 18. PMID 25788182